CLINICAL TRIAL: NCT06532487
Title: Addressing Durable Health Disparities Through Critical Time Legal Interventions in Medically Underserved Latinx and Migrant Communities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: University of Central Florida (Other); Boston University (Other); University of Puerto Rico (Other)
Responsible Party: Principal Investigator, Miguel Muñoz-Laboy, Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AWD00003786
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Health Harming Legal Needs
Keywords: medical-legal partnerships, health harming legal needs, medically underserved communities, Latinx communities, Migrant communities, FQHC

STUDY DESIGN:
Intervention Model Description: Hybrid type II effectiveness-implementation trial with a cluster randomized design.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Critical Time Medical-Legal Partnership Intervention (Experimental): Patients receiving care at an intervention health center will (a) be screened for health-harming legal needs. Those who meet eligibility criteria will be offered the opportunity to meet with a lawyer to review and explain their legal risks, rights, and remedies, (b) will be provided direct legal representation to mitigate or eliminate those legal needs, and (c) will consent to tracking of legal case management activity and outcomes and health outcomes in ways that accord with patient autonomy/consent, study expectation.
  Interventions: Other: Critical Time Medical-Legal Partnership Intervention
- Control (No Intervention): Patients receiving care at a health center in the control arm of the study in the control or "no intervention" arm of the study will (a) be screened for health-harming legal needs. Those who meet eligibility criteria will (b) be provided basic legal information and referral to legal aid, and (c) will consent to tracking of legal and health outcomes in ways that accord with patient autonomy/consent, study expectation.

INTERVENTIONS:
Other: Critical Time Medical-Legal Partnership Intervention — Utilizing a hybrid type II effectiveness-implementation trial with a cluster randomized design in six predominantly Latino-serving federally qualified health centers (FQHCs) in three major urban settings, we are examining whether integrating legal services into existing health clinics that serve Latinx and recent migrant communities can improve engagement in care and improve the health of Latinx/Hispanic and recent migrants.
  Arms: Critical Time Medical-Legal Partnership Intervention

SUMMARY:
This clinical trial will examine the effects of legal services on primary care outcomes for medically underserved communities.

The aims of the study are:

1. To test the effectiveness and cost-benefits of a critical-time intervention Medical-Legal Partnership (CTI-MLP) on patient outcomes.
2. To determine the most efficient mechanisms for CTI-MLP delivery.
3. To develop innovative community engagement strategies for addressing health-harming legal needs within community health centers.

Eligible patients will be asked to complete a questionnaire 4 times, first when they join the study and then at 3 months, 6 months, and 12 months. In the survey, they will be asked to provide information about themselves, their health care, aspects of their daily life, and hardships they face. They will also allow researchers to access their electronic health record information housed in the community-based organization and attorney notes.

Patient information will be completely confidential and de-identified, meaning, the research team will not know the identity of the person who answered the questions.

Participating community health centers will be randomized (assigned by chance) to provide basic legal information and referral to legal aid; or have an attorney on-site to provide legal aid to those who screen for legal needs.

DETAILED DESCRIPTION:
In this study, we proposed that providing legal services within primary care can enhance healthcare delivery efficiency by addressing legal needs (such as barriers to health insurance, medical treatments, housing safety, employment stability, and other legal needs) that can disrupt care to patients.

The proposed study, led by researchers at Stony Brook University, Boston University, University of Central Florida (UCF), and the University of Puerto Rico in partnership with the National Center for Medical-Legal Partnerships, UCF School of Medicine's Implementation Science Lab, and six federally qualified health centers; will precisely examine the effects of legal services on primary care outcomes for medically underserved communities. We will conduct a hybrid type II effectiveness-implementation trial with a cluster randomized design in 6 federally qualified health centers (FQHCs) in Pennsylvania, New York, and Puerto Rico to test a Critical-time Intervention Medical-Legal Partnership (CTI-MLP) approach compared to the standard of care. Three FQHCs will receive a CTI-MLP approach that includes provision of legal aid and capacity building through team-facing legal support. The other three FQHCs will receive legal education and awareness, including information about community-based legal organizations. Over a 12-month period, the team will collect (1) patients' health and functioning, including overall physical health, mental health, social health, pain, fatigue, and overall perceived quality of life; (2) data on legal needs and risk factors (3) longitudinal patient clinical outcomes (N=960); and (4) FQHC staff (N=180) and clinic-level indicators, including provider-patient communication and readiness for continued implementation and sustainability.

We will assemble a Latinx and migrant community advisory board and a scientific advisory board with medical-legal partnership expertise. Active engagement will ensure the effective translation and dissemination of our findings into practice. With new Medicaid models emerging that offer reimbursement for some social care provision, state officials can also use data to consider expansion of Medicaid services to include the coordination and provision of social and legal services. Completion of this project will result in an innovative, evidence-based intervention package to improve health outcomes for highly vulnerable communities.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included in the trial if they meet all the following criteria: 1) ages 13 or older, 2) impacted by acute health-harming legal needs or risks (confirmed by screening developed in preparation for this proposal); 3) willing and able to consent to participate in the trial (including accessing EHR at the FQHC); and, 4) do not intend to relocate within the 12 months following their enrollment in the study.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria will be excluded from the trial. Individuals who self-report having been sentenced to serve under state or federal custody, with a sentence to begin within 12 months from proposed enrollment in the study, will also be excluded from the trial.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1140 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
PROMIS Global Health-10 | 1) baseline (point of contact with patient); 2) 3-month, 3) 6- month, 4) and 12-month follow ups.
  PROMIS Global Health-10, a self-administered measured included in the survey described below. It includes general domains of health and functioning including overall physical health, mental health, social health, pain, fatigue, and overall perceived quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Betances Health Center, New York, New York, United States